CLINICAL TRIAL: NCT03282760
Title: A Phase I Multicenter Study of Allogenic, Intracerebroventricular Human Neural Stem Cells Transplantation for the Experimental Treatment of Secondary Progressive Multiple Sclerosis Patients
Brief Title: Safety Study of Human Neural Stem Cells Injections for Secondary Progressive Multiple Sclerosis Patients
Acronym: NSC-SPMS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Collaborators: Associazione Revert ONLUS (Unknown); Neurocenter of Southern Switzerland (Other); Fondazione Cellule Staminali (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NSC SPMS; 2015-004855-37 (EudraCT Number)
Record Dates: First submitted 2017-08-09; First posted 2017-09-14 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Secondary-progressive Multiple Sclerosis
Keywords: Cell Transplantation; Neural Stem Cells
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Intervention Model Description: Fifteen to 24 patients affected by SPMS will be enrolled, according to a "standard" phase I design over 18 months. All patients will enter a 3 months run in phase. Thereafter they will receive one of four different doses of allogenic hNSCs (dose A=5 millions hNSCs; dose B=10 millionshNSCs; dose C=16 millions hNSCs; dose D=24 millions hNSCs).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human Neural Stem Cells Suspension (Experimental): Intraventricular injections of Allogenic human Neural Stem Cells (hNSCs) in four different dosages (5, 10,16 or 24 millions)
  Interventions: Biological: Human Neural Stem Cells

INTERVENTIONS:
Biological: Human Neural Stem Cells — Allogenic human Neural Stem Cells (hNSCs) in four different dosages (5, 10, 16 or 24 millions). hNSCs are produced by the Laboratorio Cellule Staminali of Terni according to GMP guidelines and are obtained from brain specimens of several fetal human donors from spontaneous miscarriages occurred after the 8th week after conception.

SUMMARY:
This will be a phase I, open, multicenter, international study performed by 3 participating centres across two countries (Italy and Switzerland). Fifteen to 24 patients affected by SPMS will be enrolled, according to a "standard" phase I design over 18 months. All patients will enter a 3 months run in phase. Thereafter they will receive one of four different doses of allogenic hNSCs (dose A=5 millions hNSCs; dose B=10 millions hNSCs; dose C=16 millions hNSCs; dose D=24 millions hNSCs). Following hNSCs injection, all SPMS patients will receive immunosuppression with tacrolimus for 6 months. Patients will be clinically followed monthly for 1 year and then every 6 months for the 5 years following the study completion (possibly all life long).

MRI assessments will be performed monthly for the first 6 months and then every 3 months for 5 years following the study completion.

ELIGIBILITY:
Inclusion Criteria:

1. SPMS with progressive accumulation of disability after initial relapsing course, with or without disease activity (Lublin et al. 2014).
2. EDSS ≥ 6.5 and ≤ 8
3. EDSS progression over the 2 years prior to study start of ≥ 1.0 point for patients with EDSS =6.5 at the time of inclusion , and of ≥ 0.5 points for patients with EDSS > 6.5 at the time of inclusion
4. Age ≥ 18 and ≤ 60 years
5. Failure of best medical treatment as judged by the treating neurologist and declared absence of therapeutic alternatives

Exclusion Criteria:

1. Neurological conditions other than MS.
2. Psychiatric disorders, severe cognitive decline and personality and relational disorders.
3. History or known presence of significant systemic, infectious, oncologic or metabolic disorders.
4. Presence of any other autoimmune disease.
5. Chronic infections (HBV, HCV, HIV, tuberculosis).
6. Inability to perform MRI scans.
7. Immunomodulant/immunosuppressive treatments in the last 6 months before inclusion.
8. Current participation to other experimental studies.
9. Inability to provide informed consent.
10. Any contra-indication to lumbar puncture and the surgical procedure (e.g. use of anticoagulants)
11. Pregnancy and breast feeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2021-05-29 (Actual); Study Completion 2021-05-29 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent AE | 1 year
  To Evaluate the Feasibility, Safety and Tolerability of intracerebroventricular injection of allogenic hNSCs
Percentage of Mortality in treated patients | 1 year
  Percentage of subjects (%) with death due to procedure (mortality correlated to treatment)

SECONDARY OUTCOMES:
Change in Functional disability | Up to 1 year
  this will be measured by the change of the Expanded Disability Scale (EDSS-disability score about pyramidal, cereberral, brainstem, sensory, bowel and bladder, visual, cerebral Functional Systems) during the study period.
Change in Functional disability | Up to 1 year
  this will be measured by the change of the the Multiple Sclerosis Functional Composite (MSFC-scores about upper extremity function, ambulation and cognitive function) during the study period.
Activity of Cognitive function | Up to 1 year
  This will be measured as the mean change of the score of the RAO Brief Repeatable Battery of Neuropsychological Test, during the study period.
Relapses Rate | Up to 1 year
  Relapses will be measured by the change in EDSS scale
Relapses Rate | Up to 1 year
  Relapses will be measured by the Imaging evaluations
MS Biomarkers | Up to 1 year
  Investigation of potential candidate biomarkers able to monitor disease activity and predict clinical course in MS (Neurofilaments)
Alteration in Neurophysiological parameters | Up to 1 year
  Assessed by Evoked Potentials.

CONTACTS AND LOCATIONS:
Overall Officials: Angelo L Vescovi, PhD, Study Director — Casa Sollievo della Sofferenza IRCCS
Locations (3):
- Italy (2):
  - Casa Sollievo della Sofferenza - IRCCS, San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera Santa Maria di Terni, Terni
- Neurocentro della Svizzera Italiana, Istituto di Neurosienze cliniche della svizzera italiana, Centro sclerosi Multipla, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: CSR

REFERENCES:
- [Background] Gelati M, Profico D, Projetti-Pensi M, Muzi G, Sgaravizzi G, Vescovi AL. Culturing and expansion of "clinical grade" precursors cells from the fetal human central nervous system. Methods Mol Biol. 2013;1059:65-77. doi: 10.1007/978-1-62703-574-3_6. PMID 23934834
- [Background] Mazzini L, Gelati M, Profico DC, Sgaravizzi G, Projetti Pensi M, Muzi G, Ricciolini C, Rota Nodari L, Carletti S, Giorgi C, Spera C, Domenico F, Bersano E, Petruzzelli F, Cisari C, Maglione A, Sarnelli MF, Stecco A, Querin G, Masiero S, Cantello R, Ferrari D, Zalfa C, Binda E, Visioli A, Trombetta D, Novelli A, Torres B, Bernardini L, Carriero A, Prandi P, Servo S, Cerino A, Cima V, Gaiani A, Nasuelli N, Massara M, Glass J, Soraru G, Boulis NM, Vescovi AL. Human neural stem cell transplantation in ALS: initial results from a phase I trial. J Transl Med. 2015 Jan 27;13:17. doi: 10.1186/s12967-014-0371-2. PMID 25889343
- [Background] Pluchino S, Gritti A, Blezer E, Amadio S, Brambilla E, Borsellino G, Cossetti C, Del Carro U, Comi G, 't Hart B, Vescovi A, Martino G. Human neural stem cells ameliorate autoimmune encephalomyelitis in non-human primates. Ann Neurol. 2009 Sep;66(3):343-54. doi: 10.1002/ana.21745. PMID 19798728
- [Background] Pluchino S, Quattrini A, Brambilla E, Gritti A, Salani G, Dina G, Galli R, Del Carro U, Amadio S, Bergami A, Furlan R, Comi G, Vescovi AL, Martino G. Injection of adult neurospheres induces recovery in a chronic model of multiple sclerosis. Nature. 2003 Apr 17;422(6933):688-94. doi: 10.1038/nature01552. PMID 12700753
- [Background] Ferrari D, Zalfa C, Nodari LR, Gelati M, Carlessi L, Delia D, Vescovi AL, De Filippis L. Differential pathotropism of non-immortalized and immortalized human neural stem cell lines in a focal demyelination model. Cell Mol Life Sci. 2012 Apr;69(7):1193-210. doi: 10.1007/s00018-011-0873-5. Epub 2011 Nov 11. PMID 22076651
- [Derived] Leone MA, Gelati M, Profico DC, Gobbi C, Pravata E, Copetti M, Conti C, Abate L, Amoruso L, Apollo F, Balzano RF, Bicchi I, Carella M, Ciampini A, Colosimo C, Crociani P, D'Aloisio G, Di Viesti P, Ferrari D, Fogli D, Fontana A, Frondizi D, Grespi V, Kuhle J, Laborante A, Lombardi I, Muzi G, Paci F, Placentino G, Popolizio T, Ricciolini C, Sabatini S, Silveri G, Spera C, Stephenson D, Stipa G, Tinella E, Zarrelli M, Zecca C, Ventura Y, D'Alessandro A, Peruzzotti-Jametti L, Pluchino S, Vescovi AL. Phase I clinical trial of intracerebroventricular transplantation of allogeneic neural stem cells in people with progressive multiple sclerosis. Cell Stem Cell. 2023 Dec 7;30(12):1597-1609.e8. doi: 10.1016/j.stem.2023.11.001. Epub 2023 Nov 27. PMID 38016468
- [Derived] Gelati M, Profico DC, Ferrari D, Vescovi AL. Culturing and Expansion of "Clinical Grade" Neural Stem Cells from the Fetal Human Central Nervous System. Methods Mol Biol. 2022;2389:57-66. doi: 10.1007/978-1-0716-1783-0_5. PMID 34558001